CLINICAL TRIAL: NCT06639581
Title: Effect of 9 Doses of Dorsal Mechanical Stimulus on Volume Respiratory Measures on Healthy Preterms: a Pilot Study
Brief Title: Pilot Study to Evaluate Doses of Mechanical Stimulus on the Effectiveness of Preterm Breathing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, Paulina Toso, Clinical Professor, Pontificia Universidad Catolica de Chile
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 210406008
Record Dates: First submitted 2022-09-29; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Apnea of Prematurity; Intermittent Hypoxia
Keywords: preterm; hypoxia; medical device
MeSH Terms: conditions — Apnea; Premature Birth; Hypoxia

STUDY DESIGN:
Intervention Model Description: A baseline evaluation will be carried out and with the 9 doses of dorsal stimulation resulting from the combination of displacements of 3-5 -8 mm and 20-30-40 cycles per minute, randomized and performed by 2 operators each.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All the data is going to be registered by Rec Trial Software, anonimize and blind to everybody
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 3mm lifting stimulus (Active Comparator): Respiratory volume measures, vital signs and respiratory mechanics will be evaluated in 10 healthy preterm, by dorsal stimulation causing a displacement of 3 mm , performed by 2 operators .
  Interventions: Device: 20 per minute stimulus; Device: 30 per minute stimulus; Device: 40 per minute stimulus
- 5mm lifting stimulus (Active Comparator): Respiratory volume measures, vital signs and respiratory mechanics will be evaluated in 10 healthy preterm, by dorsal stimulation causing a displacement of 5 mm , performed by 2 operators .
  Interventions: Device: 20 per minute stimulus; Device: 30 per minute stimulus; Device: 40 per minute stimulus
- 8mm lifting stimulus (Active Comparator): Respiratory volume measures, vital signs and respiratory mechanics will be evaluated in 10 healthy preterm, by dorsal stimulation causing a displacement of 8 mm , performed by 2 operators .
  Interventions: Device: 20 per minute stimulus; Device: 30 per minute stimulus; Device: 40 per minute stimulus
- Basal (No Intervention): Respiratory volume measures, vital signs and respiratory mechanics will be evaluated in 10 healthy preterm basal- without stimulation- performed by 2 operators .

INTERVENTIONS:
Device: 20 per minute stimulus — crossover randomized mechanical dorsal stimuli -for one minute each- at 20-rates per minute
  Arms: 3mm lifting stimulus; 5mm lifting stimulus; 8mm lifting stimulus
Device: 30 per minute stimulus — crossover randomized mechanical dorsal stimuli -for one minute each- at 30 rates per minute
  Arms: 3mm lifting stimulus; 5mm lifting stimulus; 8mm lifting stimulus
Device: 40 per minute stimulus — crossover randomized mechanical dorsal stimuli -for one minute each- at 40 rates per minute
  Arms: 3mm lifting stimulus; 5mm lifting stimulus; 8mm lifting stimulus

SUMMARY:
The goal of this clinical trial is to compare, in healthy preterm babies, 9 doses of dorsal mechanical stimuli, in order to answer:

* if there is a dose of dorsal mechanical stimuli that improves the basal respiration.

Participants will be stimulated through a cotton shirt for one minute with each dose, while respiratory measures will be taken through a nasobuccal mask, slightly tightened by the investigator staff. All time, babies are going to be monitored and assessing that they are comfortable.

DETAILED DESCRIPTION:
Apnea of Prematurity (AOP) occurs in 90% of infants born at ≤34 weeks of gestation. Despite current treatments, these infants continue to experience intermittent hypoxia (IH) events, which lead to subsequent complications. Dorsal and extremity kinesthetic stimulation-commonly practiced in patients experiencing apnea-has been shown to trigger the infant's own respiratory effort. Several clinical studies have demonstrated that mechanized or reactive stimulation, performed with various devices and at different intensities, decreases the number of apneas and reduces the time spent with oxygen saturation levels below 90%, a measure of IH. However, there are also reports of no favorable effects with certain other stimulation mechanisms.

To study the kinesthetic mechanism, a pilot study was conducted on 10 healthy premature infants. The infants were dorsally stimulated using a surgical glove inflated by a mechanical ventilator at rates of 20 and 40 cycles per minute, applying a standardized stimulus independent of weight and gestational age. The main results showed that, during the stimulation period, the respiratory rate decreased by 19-50% compared to baseline (without stimulation), while oxygen saturation increased by 2-7 percentage points. Additionally, it was observed that synchronization of breathing with the dorsal stimulus occurred 0-77% of the time.

These observations could be explained by the assumption that premature infants achieved more effective breaths through stimulation, recruiting more alveolar units, and potentially triggering the Hering-Breuer reflex, which inhibits subsequent respiratory efforts. Although these findings were statistically significant based on the analysis of paired sample means, not all infants responded in the same way.

Method: A pilot study involving 10 healthy preterm infants (24-34 weeks gestational age) will be conducted. The infants will be stimulated on their backs with different combinations of lifting (3, 5, and 8 mm) and frequency (20, 30, and 40 cycles per minute) using a shirt equipped with an inflating-deflating actuator. The main outcome will be a comparison of minute ventilation and tidal volumes at baseline and with the different stimulation doses. The software "Rec Trial" will be used to record vital signs, operational settings, respiratory volumes, and patterns for repeated measures ANOVA analysis. The expected results are to find the optimal combination of lifting and frequency stimulus to optimize minute ventilation and/or detect relevant respiratory patterns that improve minute ventilation.

ELIGIBILITY:
Inclusion Criteria: 24-34 weeks of birth gestational age (BGA) preterms, healthy -

Exclusion Criteria: respiratory support, thoracic or abdominal malformations-recent surgeries, hypotonic syndromes

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Comparison of mean of Tidal Volume(TV) between the doses of dorsal mechanical stimuli | 1 minute for each intervention ( dose)
  repeated measures ANOVA for mean of Tidal Volume ( ml/kg)
Comparison of mean of Minute Ventilation (MV) between the doses of dorsal mechanical stimuli | 1 minute for each intervention ( dose)
  repeated measures ANOVA for mean of MV ( ml/kg/ min)

SECONDARY OUTCOMES:
Comparison of mean of Respiratory Rate (RR)between the doses of dorsal mechanical stimuli | 1 minute for each intervention ( dose)
  repeated measures ANOVA for mean RR (rpm)
Comparison of mean of Cardiac Rate (CR)between the doses of dorsal mechanical stimuli | 1 minute for each intervention ( dose)
  repeated measures ANOVA for mean CR (rpm)
Comparison of mean of percent of oxygen saturation (Sats) between the doses of dorsal mechanical stimuli | 1 minute for each intervention ( dose)
  repeated measures ANOVA for mean Sats (percent)

OTHER OUTCOMES:
Analyss of pattern of respiratory drive between the doses of dorsal mechanical stimuli | 1 minute for each intervention ( dose)
  Qualitative description of the respiratory drive( synchronicity-asynchronicity)
Risk manangement | 45-60 minutes each patient
  Description of Adverse Events( Neonatal Infant Pain Score (NIPS) >2-skin reactions-Apnea- Desaturation)

CONTACTS AND LOCATIONS:
Overall Officials: Paulina A Toso, MD, Study Director — Pontificia Universidad Catolica de Chile
Locations (1):
- Puc, Nicu, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No